CLINICAL TRIAL: NCT05383859
Title: Effectiveness of a Primary Care Diet and Physical Activity Educational Program for Patients With Type 2 Diabetes Mellitus
Brief Title: Diet and Physical Activity Program for Type 2 Diabetes Mellitus
Acronym: Td2Ast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Collaborators: Servicio de Salud del Principado de Asturias. Área Sanitaria III (Unknown)
Responsible Party: Principal Investigator, Rubén Martín Payo, Lecturer, Researcher, PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.014
Record Dates: First submitted 2022-03-31; First posted 2022-05-20 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): 1. Completing the consent and the pre-intervention questionnaires, anthropometric and HbA1c measurements.
  2. Dietary and/ or physical activity: face to face plus written material
  3. 3 months later: motivational phone call.
  Interventions: Behavioral: Intervention
- Control group (CG) (No Intervention): 1. Completing the consent and the pre-intervention questionnaires, anthropometric and HbA1c measurements.
  2. Usual care

INTERVENTIONS:
Behavioral: Intervention — 1. Dietary and/ or physical activity: face to face plus written material (at baseline)
  2. 3 months later: motivational phone call.
  Arms: Intervention Group (IG)

SUMMARY:
An individualized educational intervention are going to be developed. Its based on the COM-B model, designed and applied by Primary Care nursing professionals for patients with type 2 diabetes mellitus. Its expected that participants, after a 6 month intervention, face to face and telephone, will improve their adherence to healthy behaviors related to diet and physical activity, their quality of life and the glycosylated hemoglobin figures.

ELIGIBILITY:
Inclusion Criteria:

* Be cared for by one of the nurses participating in the research team
* Ability to complete the questionnaire
* Sign the informed consent
* Keep the Primary care health center during till the end of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Diet recommendations (mean) | Change from Baseline dietary recommendations at 6 months
  Compliance with dietary recommendations. We are going to use the Motiva.Diaf DM2 questionnaire. Includes 8 questions for dietary adherence. Response in dichotomous option 0 (do not follow the recommendation) or 1 (follow the recommendation). Total score range from 0 (worst dietary compliance) to 8 (best dietary compliance).
Change in Physical activity recommendations (mean) | Change from Baseline physical activity recommendations at 6 months
  Compliance with physical activity recommendations. We are going to use the Motiva.Diaf DM2 questionnaire. Includes 4 questions for physical activity recommendations. Response in dichotomous option 0 (do not follow the recommendation) or 1 (follow the recommendation). Total score range from 0 (worst dietary compliance) to 4 (best dietary compliance).
  Result: mean number of recommendations followed.

SECONDARY OUTCOMES:
Change in HbA1c (Mean percentage) | Change from Baseline % of HbA1c at 6 months
  % of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Martin, PhD, Principal Investigator — University of Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
IPD aren´t be shared